CLINICAL TRIAL: NCT06085495
Title: Clinical Comparative Study of Mechanical Thrombectomy and Simple Anticoagulation Therapy for Acute Lower Limb Deep Vein Thrombosis in Tumor Patients Under VTE Prevention and Control System
Brief Title: Mechanical Thrombectomy for Acute Lower Limb Deep Vein Thrombosis in Tumor Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y031
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cancer Patients With Acute Lower Limb Deep Vein Thrombosis (DVT)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improved approach mechanical thrombectomy (PMT) group (Other)
  Interventions: Procedure: mechanical thrombectomy (PMT)
- Traditional simple anticoagulant group (No Intervention)

INTERVENTIONS:
Procedure: mechanical thrombectomy (PMT) — After the establishment of the pathway, Angiojet (Boco, USA) was used to infuse urokinase into the blood vessels of the thrombotic segment. After waiting for 15 minutes, mechanical thrombectomy was performed. After thrombectomy, the effectiveness of thrombectomy was evaluated through angiography. For residual thrombi, repeated thrombectomy was performed, with a maximum thrombectomy volume of 480ml. After thrombectomy, antegrade angiography of the dorsal vein of the foot was performed again. If iliac vein stenosis was found to be greater than 50%, Then, Mustang balloons (Boko, USA) that match the normal blood vessel diameter are used for dilation. If the residual stenosis after dilation is greater than 30%, Wallsten stents that match the normal blood vessel diameter are inserted (Boko, USA). After all operations are completed, a dorsalis pedis venography is performed again to evaluate the thrombus burden and calculate the immediate thrombus clearance rate and thrombus clearance level.
  Arms: Improved approach mechanical thrombectomy (PMT) group

SUMMARY:
This study will conduct a prospective single blind controlled study on the clinical efficacy and safety indicators of 50 cancer patients with acute lower limb deep vein thrombosis (DVT). The patients were randomly divided into an experimental group (improved mechanical thrombectomy (PMT) group) and a control group (traditional simple anticoagulation group) using the "envelope method", with 25 cases each. After the end of treatment, clinical prognosis evaluations were conducted on the patient's vital signs, symptoms and signs, lower limb Doppler ultrasound examination, patient PTS score (Villalta score), quality of life score (QOL), etc. at 3, 6, and 12 months. Adverse events, the presence or absence of thrombus recurrence, and re surgical intervention were recorded. This study is expected to propose a new strategy for the treatment of acute DVT in cancer patients, thereby improving the overall level of VTE prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Between the ages of 18 and 75; 2) Suffering from acute lower limb deep vein thrombosis (DVT) with a duration of less than 14 days from onset; 3) Thrombosis involving the iliac vein, femoral vein, or popliteal vein; 4) The patient has been diagnosed with tumors, including benign or malignant tumors, including surgical or conservative treatment; 5) Sign an informed consent form.

Exclusion Criteria:

* 1) Patients with a history of deep vein thrombosis of the same lower limb in the past; 2) Patients with plasma Cr levels greater than 180umol/L; 3) Patients with contraindications to thrombolytic drugs; 4) Patients with concomitant inferior vena cava thrombosis or simple calf intermuscular vein thrombosis; 5) Patients who are known to be allergic to heparin, low molecular weight heparin, contrast agents, etc; 6) Patients who have participated in clinical trials of drugs or other medical devices that interfere with this clinical trial within the past 3 months; 7) Pregnant and lactating women; 8) Patients with a life expectancy of less than 6 months, or those with other diseases that may cause difficulty in testing or significantly shorten the patient's life expectancy (<1 year), including severe liver disease, cardiac insufficiency, etc; 9) Patients with autoimmune thrombotic disease; 10) Patients who are unable or unwilling to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
The incidence of PTS at 12 months after surgery | 1 year
  Villalta Rating at 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No